CLINICAL TRIAL: NCT03974958
Title: Circulating microRNAs and Degenerative Abdominal Aorta Aneurysm: Diagnostic Specificity and Prognostic Value in Clinical Practice
Brief Title: Circulating microRNAs and Degenerative Abdominal Aorta Aneurysm
Acronym: ACTA-miRNA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2018-12
Record Dates: First submitted 2019-06-03; First posted 2019-06-05 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Abdominal Aorta Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AAA patients (Experimental): Patients with abdominal aortic aneurysm (AAA)
  Interventions: Genetic: Tissue-library
- PAOD patients (Experimental): patients with peripheral arterial obstructive disease (PAOD)
  Interventions: Genetic: Tissue-library

INTERVENTIONS:
Genetic: Tissue-library — circulating biomarkers (miRNA panel) analysis of blood samples

SUMMARY:
Abdominal aortic aneurysm (AAA) is an aortic dilatation superior or equal to 30 mm with an estimated prevalence at 8% in men over 65 year-old. It evolves with no clinical signal until the rupture of the aortic wall with dramatic outcomes. The pathophysiological mechanisms include extracellular matrix remodeling, smooth muscle cells apoptosis, aggregation and activation of inflammatory cells in the aortic wall and heredity. The initiating and regulatory processes are complex and not fully elucidated. They encompass local aortic environment (flux, thrombus, wall shear stress, pressure and adipose tissue) and patient-dependent genetic (de)regulation.

This project follows the previous prospective ACTA study that aimed at identifying clinical criteria, circulating biomarkers or imaging data for thoracic aneurysm prognosis in an AAA population. The preliminary results showed that 1) a low wall shear stress index and the luminal volume are more predictive values for a rapid AAA growth and an intraluminal thrombus than the maximal aortic diameter 2) three thoracic aortic phenotypes (normal, dilated, aneurysmal) stratify the disease extent 3) the age and the female gender are associated to an extended disease. During this study we created a biobank in which blood samples of AAA patients were collected at the time of their inclusion (T1). This new ACTA-miRNA study aims at correlating circulating biomarkers to the anatomical and biomechanical markers previously highlighted for a rapid aneurysmal growth. Circulating miRNA are involved in parietal remodeling and constitute promising targets for estimating patients-specific aortic risk.

From the literature, we thus selected 18 miRNA described to be involved in AAA biology: inflammation, remodeling, cellular homeostasis and wall shear stress. As control, we select non-AAA patients presenting with peripheral arterial obstructive disease (PAOD) matched in age, BMI, tobacco consumption, diabetes, cholesterol level and blood pressure with AAA patients enrolled in the ACTA study. During their follow-up, these ACTA patients are solicited to continue the program research and can participate to the ACTA-miRNA study. A third time analysis is performed for them (T3): we collect imaging data of total aorta required by their standard follow-up, as well as a blood sample. Differential analysis of the miRNA panel will be conducted between 1) AAA patients (T1) vs PAOD patients 2) fast-growing AAA vs slow-growing AAA 3) AAA & AAT patient group vs AAA alone and/or AAA & dilatation of thoracic aorta. 110 patients from the ACTA study are eligible to be included into the ACTA mi-RNA study. Inclusion of PAOD controls will be conducted until the number of 165 cases is reached (1:1.5 ratio).

Our primary objective is to validate a circulating-miRNA signature specific for abdominal aortic aneurysm.

ELIGIBILITY:
Inclusion Criteria:

• Case AAA T3 : Patients included in the ACTA study. They benefited from aortic imaging assessment at times T1 and T2 and were not operated on AAA.

• AOMI Case Control : Patients referred for hospitalization or referred to vascular surgery for management of chronic peripheral claudication on AOMI not associated with aneuric aneurysm evolutionary or previously operated. They must benefit from a CT angiography of the aorta and lower extremity arteries as well as a cardiac ultrasound scan.

Exclusion Criteria:

* minor patients;
* pregnant women;
* patients with cancer at the time of inclusion;
* contraindication to iodinated contrast medium: allergy to iodine, severe renal insufficiency (≤40 ml / min);
* patients presenting one of the following pathologies associated with a disruption of the activation of coagulation and / or inflammation (less than 6 weeks old):

  * Arterial thrombotic disease: acute coronary syndrome, TIA/CVD, peripheral artery acute ischemia and/or anti-vitamin K (AVK) treatment;
  * venous thrombotic pathology: peripheral venous thrombosis of less than 3 months and/or under AVK treatment, pulmonary embolism less than 6 months old and/or under AVK treatment;
  * surgery;
  * revascularization with angioplasty;
  * critical ischemia patente;
  * permanent atrial fibrillation due to associated microparticle elevation, and AVK treatment;
  * major haemorrhage;
  * acute infection.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2022-03-21 (Actual); Study Completion 2022-03-21 (Actual)

PRIMARY OUTCOMES:
Comparison of AAA miRNAs vs AOMI miRNAs | 24 months
  Analyze the diagnostic value of the 18 selected microRNAs circulating profile in degenerative aneurysmal aortic remodeling (patients with an abdominal aortic aneurysm (AAA)) in comparison with the circulating profile of the same 18 microRNAs panel in the atherosclerosis remodeling (patients with peripheral arterial occlusive disease (AOMI) without AAA)

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Garrido Pradalié, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France